CLINICAL TRIAL: NCT01873040
Title: Randomized Intervention Trial to Evaluate a Vaccine Social Media Website
Brief Title: Vaccine Social Media Randomized Intervention Trial
Acronym: VSMRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HS021492-01 (AHRQ)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Communicable Diseases
Keywords: Social Media; Vaccine; Immunization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Social media plus information pages (Experimental): Participants will have access to the vaccine social media website with information pages and social media features including discussion forums, blogs, chat with an expert, and ask an expert.
  Interventions: Behavioral: Social Media plus information pages
- Information Pages (Experimental): Participants will have website access to vaccine information pages.
  Interventions: Behavioral: Vaccine Information Pages
- Usual Care (No Intervention): Participants will not have access to the vaccine website. They will receive pediatric care as usual.

INTERVENTIONS:
Behavioral: Social Media plus information pages — Participants will receive access to the study vaccine website information pages and social media feature including blogs, discussion forums, expert chats, and ask an expert.
  Arms: Social media plus information pages
Behavioral: Vaccine Information Pages — Participants will receive access to the study vaccine website information pages.
  Arms: Information Pages

SUMMARY:
This study will assess the effectiveness of social media website devoted to vaccines to change immunization knowledge, perceptions and behavior. If effective, this intervention will represent an innovative, low cost and broadly applicable resource to reduce parental vaccination concerns.

The study has two hypothesis:

1. Parents receiving usual care plus social media website will demonstrate higher early childhood immunization rates to parents receiving either usual plus non interactive website or usual care only.
2. Parents receiving usual care plus social media website will demonstrate positive changes in knowledge, attitudes and beliefs supporting vaccination compared to parents receiving either usual care plus non-interactive website or usual care only.

DETAILED DESCRIPTION:
Participants will be enrolled in the study, stratified based on hesitancy and randomly assigned to 1 of 3 study arms and followed for 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Women >20 weeks Pregnant (including parents of children up to 1 year of age).
* >18 years of age

Exclusion Criteria:

* Non english speak
* Do not intend to use Kaiser insurance for the child

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1675 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Days under-immunized | 2 years
  Days under-immunized is a metric to identify immunization delay. For each vaccine dose calculate the difference between when the vaccine dose was actually administered and when the vaccine dose should have been administered according to the Advisory Committee on Immunization Practices (ACIP) schedule. That difference is summed across all doses and vaccines for a total number of days under-immunized for each child. Total days under immunized was calculated 200 days after life or after enrollment. If someone had 0 days at that time they were considered "up to date".

SECONDARY OUTCOMES:
Knowledge, Attitudes and Beliefs about immunizations | Baseline, Child age 3-5 months, Child age 12-15 months
  Knowledge, attitudes, and beliefs will be measured with a survey at up to 3 time points during the study: 1) Initial enrollment in the study, 2) child's ag=4-6 months and 3) child's age=11-13 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Glanz, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Colorado Institute for Health Research, Denver, Colorado, United States

REFERENCES:
- [Derived] O'Leary ST, Narwaney KJ, Wagner NM, Kraus CR, Omer SB, Glanz JM. Efficacy of a Web-Based Intervention to Increase Uptake of Maternal Vaccines: An RCT. Am J Prev Med. 2019 Oct;57(4):e125-e133. doi: 10.1016/j.amepre.2019.05.018. Epub 2019 Aug 27. PMID 31471001
- [Derived] Daley MF, Narwaney KJ, Shoup JA, Wagner NM, Glanz JM. Addressing Parents' Vaccine Concerns: A Randomized Trial of a Social Media Intervention. Am J Prev Med. 2018 Jul;55(1):44-54. doi: 10.1016/j.amepre.2018.04.010. Epub 2018 May 14. PMID 29773490